CLINICAL TRIAL: NCT00535964
Title: Anxiety Sensitivity, Tobacco Use, and Panic Among Adolescents
Brief Title: Evaluating the Relationship Between Tobacco Use, Anxiety Sensitivity, and Panic in Adolescents
Status: Completed | Type: Observational
Sponsor: University of Arkansas, Fayetteville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ellen Leen-Feldner, Professor of Psychology, University of Arkansas, Fayetteville
Other Study IDs: R03MH077692 (NIH); R03MH077692 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Panic Disorder
Keywords: Cigarette Smoking; Tobacco Use; Adolescents; Anxiety Sensitivity (AS)
MeSH Terms: conditions — Panic Disorder; Cigarette Smoking; Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Psychologically healthy adolescents, evenly divided across the various stages of smoking uptake

SUMMARY:
This study will determine whether there is a relationship between tobacco use and a heightened response to panic-producing events among adolescents. This study is fundamental research. It was not a Clinical Trial.

DETAILED DESCRIPTION:
Growing up is hard enough, and adolescence can be a particularly stressful time in people's lives as they adjust to the transition from childhood to adulthood. Peer pressure can add to this anxiety, making it more likely for teens to take part in risky behaviors such as smoking cigarettes. Every day, more than 4,000 teens smoke their first cigarette and nearly half of those teens will become regular, daily smokers. Cigarette smoking is associated with a multitude of health risks, including an increased likelihood of experiencing panic attacks, anxiety disorders, and depression. This study will evaluate a group of teens, ranging from those who have never smoked to those who smoke daily, to determine whether there is a relation between adolescent smoking history and their vulnerability to panic-producing situations.

Participants in this study will undergo a brief medical screening, followed by a short interview that will include several questionnaires regarding emotions, experiences, and personal habits. Participants will then attend a series of laboratory assessments for 1 hour. The first assessment will include a 3-minute voluntary hyperventilation procedure in which participants will be directed when to breathe in and when to breathe out, at a faster rate than normal. Participants will then take part in two computerized tasks: one will be a computerized task that involves blowing up a balloon and deciding when to quit before the balloon pops; the other task will involve choosing hypothetical amounts of money now or after a period of delay. During the laboratory assessments, all participants will have electrodes attached to their bodies and sensors around their chests to measure heart rate, palm sweating, and muscle tension. Results from this study will be used to evaluate the association between smoking and increased panic levels under stressful conditions among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents, ranging from those who have never smoked to those who smoke daily

Exclusion Criteria:

* Current or past diagnosis of a panic disorder
* Acute or chronic cardiopulmonary or respiratory illness (e.g., asthma or bronchitis)
* Pregnant

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be 180 psychologically healthy adolescents, evenly divided across the various stages of smoking uptake (i.e., non-smokers, tried smoking, experimenters, regular smokers, and daily smokers).
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Relationship between cigarette smoking and panic vulnerability | Measured at completion of laboratory testing analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W. Leen-Feldner, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States